CLINICAL TRIAL: NCT04591782
Title: Exploratory Study to Determine the Bioavailability of Sugar From Pomegranate Juice (PJ) vs. Sucrose
Brief Title: Investigation of PJ vs. Sugar on Glucose Levels in Healthy and Prediabetic Subjects
Acronym: PSW
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Zhaoping Li, Chief / Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 18-001720
Record Dates: First submitted 2020-10-02; First posted 2020-10-19 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Diabete Type 2; Pre Diabetes
Keywords: pomegranate; antioxidants; prediabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Glucose Intolerance; Prediabetic State | interventions — Water

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- PomJuice (PJ) (Experimental): 8 oz of PJ
  Interventions: Other: PomJuice
- Sugar Water (Active Comparator): 8 oz of water with 18.6 g of glucose + 18.3 g of fructose dissolved into it
  Interventions: Other: Sugar Water
- Water (Other): 8 oz of water
  Interventions: Other: Water

INTERVENTIONS:
Other: PomJuice — Drink 8 oz pomegranate juice
  Arms: PomJuice (PJ)
Other: Water — Drink 8 oz water
  Arms: Water
Other: Sugar Water — Drink 8 oz of water with 18.6 g of glucose + 18.3 g of fructose dissolved in
  Arms: Sugar Water

SUMMARY:
Pomegranate fruits and products, including juice, tea, wine and extracts are widely consumed and recognized for their health benefits. Pomegranate fruit possesses strong antioxidant, anti-inflammatory and antiproliferative properties. The effects of pomegranate on type 2 diabetic (T2DM) conditions have previously been reported. Although 8 oz. of Pom juice (PJ) contains 36.9 g of sugar, 12-week PomJ supplementation did not change plasma advanced glycated end-products, fasting glucose and HbA1C, but reduced lipid peroxidation in T2D subjects. Additionally, acute PJ consumption has been shown to lower postprandial glycemic response of a meal with high glycemic index (GI) and lower fasting blood glucose, and long-term PomJ consumption did not worsen diabetic markers. However, a large knowledge gap still exists regarding the form of sugars in PJ and the hormonal responses to PJ consumption in different physiological conditions. Therefore currently the consumption of PJ is not recommended for individuals with T2DM. This clinical study will focus on the short-term effects of PJ consumption on different diabetic variables to further evaluate the health benefits of PJ for T2DM.

DETAILED DESCRIPTION:
This study aims to measure the effects of PJ vs. sugar on glucose and insulin levels in apparently healthy normal weight and prediabetic overweight and obese subjects. Participants will be asked to consume one serving of PJ, sugar mix and water separated by one week of beige diet without PJ consumption (crossover design). The PJ will be provided by POMWonderful. Timed blood collections over a three-hour period following the juice/sugar/water consumption will be used to measure how PJ vs. sugar mix vs. water affects glucose metabolism/insulin sensitivity in human subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age 20-50 years and any racial/ethnic group
2. Typically consume low fiber/polyphenol diet (beige diet)
3. Healthy, normal weight individuals with a BMI of >18 to 26.9 kg/ m2 with fasting serum glucose <100mg/dL or A1c <5.7
4. Prediabetic, obese individuals with a BMI of >27 kg/ m2 and fasting serum glucose >100, but <126 mg/dL or A1c >5.7% but < 6.4%]
5. Subjects must read and sign the informed consent prior to participation
6. Subjects must be in generally good health
7. Subjects must be able and willing to comply with the requirements of the protocol.

Exclusion Criteria:

1. Eating a high fiber/polyphenol diet or taking any medication or dietary supplements that interfere with the absorption of polyphenols.
2. History of gastrointestinal surgery, diabetes mellitus on medications, or other serious medical condition, such as chronic hepatic or renal disease, bleeding disorder, congestive heart disease, chronic diarrhea disorders, myocardial infarction, coronary artery bypass graft, angioplasty within 6 months prior to screening, current diagnosis of uncontrolled hypertension (defined as systolic BP >160mmHg, diastolic BP > 95mmHg), active or chronic gastrointestinal disorders, bulimia, anorexia, laxative abuse, or endocrine diseases (except thyroid disease requiring medication) as indicated by medical history
3. Any subject currently taking blood thinning medications such as Warfarin or Coumadin
4. Currently uses tobacco products.
5. Currently has an alcohol intake > 20 g ⁄ day;
6. Currently has a coffee intake > 3 cups ⁄ day;
7. Screening laboratory value outside of the laboratory normal range that is considered clinically significant for study participation by the investigator.
8. Using prebiotics, probiotics, yogurt, and/or any fiber supplements regularly
9. Allergy or sensitivity to pomegranate. Subjects will be excluded if there is a prior history of such sensitivity. Since these foods are commonly eaten and allergies are rare, subjects should be aware of this sensitivity prior to entering the study. In addition, any subject with a history of allergy or anaphylaxis of any kind will be excluded
10. Taking antibiotics or laxatives within the past 3 months
11. Is unable or unwilling to comply with the study protocol.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2019-02-01 (Actual); Primary Completion 2021-12-20 (Actual); Study Completion 2021-12-20 (Actual)

PRIMARY OUTCOMES:
Number of participants with acute response to sugar water vs. pom juice vs. water | 2 hours
  Compare the difference in blood glucose response to consuming PomJ compared to the same amount of sugar (fructose and glucose) mixed in water in a cross over study design
Number of participants with hormonal changes in response to sugar water vs. pom juice vs. water | 15 days
  Compare the plasma concentration of principle hormones involved in glucose regulation (insulin, C-peptide, glucagon) , gut hormones (GLP-1 and GIP) and triglycerides.
Number of participants with acute response of plasma nitric oxide (NO) from sugar water vs. pom juice vs. water | 2 hours
  Compare the acute response of plasma nitric oxide (NO) in participants who consume sugar alone, water alone or pomegranate juice
Impact of gut microbiome in glycemic response to pom juice vs. sugar water | 15 days
  Compare the glycemic response and the ability to form microbiote urolithin from pomegranate ellagatanins in participants who consume pom juice vs. water.

CONTACTS AND LOCATIONS:
Overall Officials: Zhaoping Li, MD, PhD, Principal Investigator — UCLA Professor of Medicine
Locations (1):
- UCLA Center for Human Nutrition, 1000 Veteran Ave., Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: Undecided